CLINICAL TRIAL: NCT06300112
Title: The Effect of Pregnancy Yoga on Perceived Stress, Quality of Sexual Life and Sleep Level
Brief Title: Prenatal Yoga on Stress, Quality of Sexual Life and Sleep Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Emine Akca, Assist. Prof. Dr. in the Amasya University Midwifery Department, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya Univ_emine.akca
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stress; Sexuality; Sleep
Keywords: Midwifery; Perceived Stress; Sexual Quality of Life; Sleep; Pregnancy
MeSH Terms: conditions — Sexuality | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: A randomized-controlled trial with pretest-posttest control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Yoga
  Interventions: Behavioral: YOGA
- Control group (No Intervention): No Intervention

INTERVENTIONS:
Behavioral: YOGA — Yoga will be applied to the experimental group for a total of 12 sessions, two sessions per week (90 minutes) for six weeks.
  Arms: Experimental group

SUMMARY:
The study will investigate the effects of pregnancy yoga on perceived stress, quality of sexual life and sleep level. A total of 100 pregnant women are planned to be included in the study. Data will be collected with the "Personal Information Form", "Perceived Stress Scale" and "Sexual Quality of Life Questionnaire-Female". Yoga will be applied to the experimental group for a total of 12 sessions, two sessions per week (90 minutes) for six weeks. The research predicts that yoga will reduce the stress perceived by pregnant women, increase the quality of sexual life and positively affect sleep patterns.

DETAILED DESCRIPTION:
Although pregnancy is a natural process, the change in physiological and psychosocial balance and the differentiation of roles in life require bio-psychosocial adaptation for the pregnant woman and her environment. In addition to strengthening the uterine and perineal muscles and supporting the spine, yoga is effective in dealing with common problems of pregnancy such as poor blood circulation, blood pressure fluctuations, excessive weight gain, fatigue, edema and urinary problems. The study will investigate the effects of pregnancy yoga on perceived stress, quality of sexual life and sleep level. A total of 100 pregnant women are planned to be included in the study. Data will be collected with the "Personal Information Form", "Perceived Stress Scale" and "Sexual Quality of Life Questionnaire-Female". Yoga will be applied to the experimental group for a total of 12 sessions, two sessions per week (90 minutes) for six weeks. The research predicts that yoga will reduce the stress perceived by pregnant women, increase the quality of sexual life and positively affect sleep patterns.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy week between 24 and 34,
* Able to read and write Turkish,
* No communication problems,
* Those who voluntarily agreed to participate in the research

Exclusion Criteria:

* Those who have risky pregnancies,
* Those with diagnosed psychiatric problems,
* Participating in a different training program (meditation, relaxation, etc.)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived stress level | 6 weeks
  This will be measured using "Perceived Stress Scale". The minimum score that can be obtained from the scale is "0", the maximum score is "32", and as the scale score increases, perceived stress level also increase.
Sexual Quality of Life | 6 weeks
  This will be measured using "Sexual Quality of Life Questionnaire-Female". The minimum score that can be obtained from the scale is "18", the maximum score is "108". The total score obtained from the scale must be converted to 100. As the scale score increases, perceived stress level also increase.

OTHER OUTCOMES:
Sleep patterns | 6 weeks
  Participants' sleep patterns will not be evaluated with a scale. Therefore, it does not have a specific scoring. The sleep patterns of the participants will be evaluated with questions created by the researchers.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İbici Akça, Principal Investigator — Amasya University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No